CLINICAL TRIAL: NCT04596943
Title: [68Ga]Ga-DOTA-(RGD)2 PET/CT Imaging of Activated Endothelium in Lung Parenchyma of COVID-19 Patients
Brief Title: RGD PET/CT Imaging in COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL73551.091.20; 2020-001325-31 (EudraCT Number)
Record Dates: First submitted 2020-10-20; First posted 2020-10-22 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Endothelial Dysfunction; PET Imaging
Keywords: COVID-19; endothelial dysfunction; PET imaging; RGD-peptides
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: [68Ga]Ga-DOTA-(RGD)2 PET/CT — We have developed a dimeric cyclic RGD peptide conjugated with DOTA as a chelator. If labeled with the positron emitting radionuclide Gallium-68 (68Ga), [68Ga]Ga-DOTA-(RGD)2 can be used to visualize αvβ3 integrin expression with PET
  Other Names: RGD-PET/CT

SUMMARY:
Aim: We aim to evaluate αvβ3 integrin expression in proven COVID-19 infected patients with indicative findings on routine contrast-enhanced CT using [68Ga]Ga-DOTA-(RGD)2. If activated vascular endothelium in the lung parenchyma proceeds ARDS, as frequently observed during COVID-19 infection, imaging αvβ3 integrin expression using PET/CT could have potential as a clinical tool to characterize patients at early stages during disease and guide development of novel treatments targeting the vascular endothelium.

Study design: This is a prospective, observational non-randomized pilot study. Maximum 10 patients will undergo a [68Ga]Ga-DOTA-(RGD)2 PET/CT scan and CT-subtraction scan in the same procedure. 10-minutes/bed position static [68Ga]Ga-DOTA-(RGD)2 PET/CT scans of the thorax will be acquired starting at 60 minutes post injection.

Study population: Maximum 10 patients from the Infectious Diseases ward with proven COVID-19 infection and indicative pulmonary abnormalities on contrast-enhanced CT (CORADS 4-5) undergo PET/CT scans after injection of 70 μg (200 MBq) [68Ga]Ga-DOTA-(RGD)2 and CT-subtraction.

Intervention: All patients will undergo a [68Ga]Ga-DOTA-(RGD)2 PET/CT scan, and in the same procedure, a CT-subtraction scan.

Primary study objective: The primary objective of this study is to demonstrate and quantitate activation of the endothelium in the lung vasculature using [68Ga]Ga-DOTA-(RGD)2 PET/CT.

Secondary study objectives:

1. To assess the spatial correlation between [68Ga]Ga-DOTA-(RGD)2 uptake and abnormal findings on routine contrast-enhanced CT scan of the chest
2. To assess the spatial correlation between [68Ga]Ga-DOTA-(RGD)2 and CTS of the lung parenchyma
3. To assess the correlation between [68Ga]Ga-DOTA-(RGD)2 and laboratory results
4. To explore the correlation between [68Ga]Ga-DOTA-(RGD)2 uptake and clinical course of disease

ELIGIBILITY:
Inclusion Criteria:

* a microbiologically proven SARS-CoV-19 infection
* pulmonary involvement as demonstrated on recent (<1 week) chest CT, classified as CORADS 4 or 5, with indicative findings such as ill-demarcated multifocal ground glass opacities, mixed ground glass and consolidations, predominant peripheral and basal distribution, vascular thickening, round shaped and/or (reversed) halo
* More than or equal to 18 years of age;
* Ability to provide written informed consent.

Exclusion Criteria:

• Contra-indication for PET: Pregnancy; Breast-feeding; Severe claustrophobia.

* Contra-indication for administration of iodine-containing contrast agents.
* Saturation <94% at room air (without need of additional oxygen)
* Previously documented lung abnormalities that can interfere with interpretation of research scans, e.g. extensive fibrosis, known interstitial lung disease, pulmonary metastases, known pulmonary involvement of granulomatous diseases.
* Oth Estimated creatinine clearance < 30mL/min according to the Cockcroft-Gault formula (or local institutional standard method) OR oligo-uric patients (<400mL/24hr)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for this pilot study exists of 10 evaluable patients with a proven SARS-CoV-19 infection and pulmonary involvement as demonstrated on chest CT, admitted to the Infectious Diseases ward. Patients presenting in the Radboud University Medical Center will be considered for recruitment, if they are over the age of 18.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
uptake of [68Ga]Ga-DOTA-(RGD)2 in the lung parenchyma | 2 months
  The main study parameter is the uptake of [68Ga]Ga-DOTA-(RGD)2 in the lung parenchyma as quantified by PET/CT (SUVmean ±SD, SUVmax ±SD and SUVpeak ±SD).

SECONDARY OUTCOMES:
spatial correlation with chest-CT | 2 months
  spatial correlation (per lung segment) with ground-glass opacities, consolidation and vascular thickening
spatial correlation with CT-subtraction | 2 months
  spatial correlation (per lung segment) with perfusion abnormalities as measured by CT-subtraction
quantitative correlation with laboratory results | 2 months
  quantitative correlation with blood counts and differentiation, ferritin, D-dimer, CRP, liver enzyme panel (ALAT, ASAT, direct and indirect bilirubin, alkaline phosphatase, gamma-GT, LDH)
explore correlation with clinical parameters | 2 months
  correlation with the following clinical parameters: (time to) eventual ICU admission, length of ICU stay (days), mechanical ventilation parameters, oxygen demand, total length of hospital stay (days)

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Genugten EAJ, van Lith TJ, van den Heuvel FMA, van Steenis JL, Ten Heggeler RM, Brink M, Rodwell L, Meijer FJA, Lobeek D, Hagmolen Of Ten Have W, van de Veerdonk FL, Netea MG, Prokop M, Nijveldt R, Tuladhar AM, Aarntzen EHJG. Gallium-68 labelled RGD PET/CT imaging of endothelial activation in COVID-19 patients. Sci Rep. 2023 Jul 17;13(1):11507. doi: 10.1038/s41598-023-37390-9. PMID 37460572